Version: Second.

Code of study: REST-ECL-2023-08

Comitè d'Ètica d'Investigació amb medicaments



## **Informed Consent Form**

| Date of presentation: 15/07/2023 |
|---|
| Main Researcher: Dra. Marta Valles. |
| Secondary researcher: Ricardo David Palacios Bañuelos, Gonzalo Blasi, |
| Kareem Istwany. |
| Tutor: Alvaro Blasi |
| Department: Restorative Dentistry |
| Research line: Basic research in dentistry |
| Research title: "Clinical and anatomical factors influencing accuracy in fully |
| guided implant placement." |
| <ul> <li>I have received verbal information about the study, and I have read the attached written information, of which I have been given a copy.</li> <li>I have understood what has been explained to me.</li> <li>I have been able to discuss the study and ask questions to the responsible professional.</li> <li>I give my consent to participate in the study and understand that my participation is entirely voluntary.</li> <li>I understand that I can withdraw at any time without affecting my future medical care.</li> <li>By signing this informed consent form, I give consent for my personal data to be used as described in this consent form, in accordance with the provisions of Organic Law 3/2018, of December 5, on the Protection of Personal Data.</li> <li>I understand that I will receive a copy of this informed consent form.</li> </ul> |
| Patient sign Date ID number: |

Universitat Internacional de Catalunya

Comitè d'Ètica d'Investigació amb medicaments



## **INVESTIGATOR'S STATEMENT**

The patient signing this consent form has received from the professional, detailed information both orally and in writing regarding the process and nature of this research study. They have had the opportunity to ask any questions regarding the nature, risks, and benefits of their participation in this study.

Main researcher sign

Date:

Name: Dra. Marta Vallés